CLINICAL TRIAL: NCT00422578
Title: Effect of Tadalafil on the Quality of Life and Sexual Life in Erectile Dysfunction (ED) Patients Previously Treated With Other Oral ED Therapy
Brief Title: Effect of Tadalafil on the Quality of Life and Sexual Life in Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9113; H6D-HL-LVGD
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Impotence; Erectile Dysfunction
Keywords: erectile dysfunction; tadalafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

INTERVENTIONS:
Drug: tadalafil
  Other Names: LY450190; Cialis; IC351

SUMMARY:
Study is a clinical study assessing the effect of oral tadalafil 10mg or 20 mg on psychosocial aspects and quality of life of erectile dysfunction patients and to compare tadalafil with previous oral erectile dysfunction medication. Study period is 13 weeks. Study patients fill in quality of life questionnaires and treatment satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* have a history of erectile dysfunction (defined as a consistent change in the quality of erection that adversely affects the patient's satisfaction with sexual intercourse)of at least 3 months duration
* have been using any oral prescription medication,but not tadalafil, for erectile dysfunction for a minimum period of 3 months before visit 1
* have responded to previous erectile dysfunction medication as assessed by the investigator

Exclusion Criteria:

* exhibit evidence of clinically significant hepatobiliary disease (including jaundice) at visit 1
* cardiovascular exclusion criteria: history of chronic stable angina treated with nitrates, recent acute cardiovascular events or procedures (myocardial infarction, coronary interventions, stroke, etc.), history of other serious cardiovascular events (e.g. arrhythmias, sudden cardiac arrest, congestive heart failure, etc.), systolic blood pressure <90mmHg or diastolic blood pressure <50mmHg at screening
* receiving treatment with cancer chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
On-demand therapy with tadalafil, as measured by the spontaneity domain of the PAIRS questionnaire increases the possibility to spontaneous sexual activity in ED patients compared with any other previous oral ED treatment.

SECONDARY OUTCOMES:
Estimate the level of quality of life (15D and LiSat-11)in treated ED patients in order to be able to compare it with existing data of the general population and patients suffering from other diseases and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere, Finland

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com